CLINICAL TRIAL: NCT05958602
Title: Improving Recruitment and Retention for Diabetes Self-Management Education and Support by Bridging Clinical-Community Linkages and Supplemental Diabetes Education Technology: A Socio-Ecological Approach
Brief Title: Improving Recruitment and Retention for Diabetes Self-Management Education and Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MedsPLUS Consulting (Other)
Collaborators: Lister Hill Center for Health Policy (Unknown); Jenkins Public Health Consulting LLC (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DSMESPilot2024; RFA-DK-20-032 (Other: National Institutes of Health)
Record Dates: First submitted 2023-06-22; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
Keywords: community health worker; dsmes; diabetes self-management education and support; Jefferson County, Alabama; diabetes technology; A1C; diabetes; stakeholder engagement; SDoH
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Technology (Experimental): The interventional group will receive a standard, evidence-based DSMES curriculum and supplemental diabetes education-related technology to assess an improvement in participation, retention, engagement, and clinical outcomes (HbA1C).
  Interventions: Behavioral: Technology
- Standard DSMES Only (Active Comparator): The control group will receive a standard, evidence-based DSMES curriculum only to assess an improvement in participation, retention, engagement and clinical outcomes (HbA1C)
  Interventions: Behavioral: Standard DSMES Only
- Traditional DSMES Recruitment Methods (Active Comparator): The traditional DSMES recruitment method participants will be recruited using traditional methods such as flyers, word of mouth, and media ads to assess the effectiveness of traditional methods on recruiting and enrollment into to pharmacist-led DSMES programs.
  Interventions: Behavioral: Traditional Recruitment Methods
- CHW-Led DSMES Recruitment Methods (Experimental): The CHW-led DSMES recruitment model participants will be recruited utilizing a CHW-led, multidirectional recruitment process involving community health workers (CHWs), primary care physicians, and community pharmacists to assess the effectiveness of a multidirectional recruitment process into pharmacist-led DSMES programs.
  Interventions: Behavioral: CHW-Led Recruitment Methods

INTERVENTIONS:
Behavioral: Technology — See previous response.
  Arms: Technology
Behavioral: Standard DSMES Only — See previous response.
  Arms: Standard DSMES Only
Behavioral: Traditional Recruitment Methods — See previous response.
  Arms: Traditional DSMES Recruitment Methods
Behavioral: CHW-Led Recruitment Methods — See previous response.
  Arms: CHW-Led DSMES Recruitment Methods

SUMMARY:
This randomized clinical trial aims to examine the effectiveness of utilizing CHWs (community health workers) and supplemental diabetes education technology to improve DSMES (diabetes self-management education and support) participation, retention, engagement, and clinical outcomes in adults in Jefferson County, AL living with diabetes. The main questions this study aims to answer are as follows:

1) Is the utilization of a multi-directional recruitment model via partnerships with community health workers and local primary care providers versus traditional recruitment methods (including using flyers, word of mouth, and media ads) effective in increasing recruitment and retention of people living with diabetes into a pharmacist-led DSMES program? 2) Is the utilization of the HICO Health Mobile application and provider dashboard as a supplementary tool alongside a standard DSMES curriculum effective at improving patient participation, retention, engagement, and clinical outcomes in a pharmacist-led DSMES program versus standard DSMES alone in Jefferson County, AL? After eligibility screenings and enrollment, participants will be randomized into two groups: one group will receive standard DSMES programming based on the 7 Self Care Behaviors and one group will receive standard DSMES programming and access to HICO Health, a diabetes-related mobile health application. The study team plans to evaluate whether a CHW- recruitment strategy will lead to an increase in referral and enrollment and whether incorporating the HICO Health application will lead to better retention, engagement, and clinical outcomes in terms of HbA1C levels.

This novel project will utilize continued stakeholder engagement, community health workers, and diabetes-related technology which we hope will increase the uptake and retention of participants in DSMES in Jefferson County, AL.

DETAILED DESCRIPTION:
Diabetes is of increasing public health concern in Alabama due to high prevalence, incidence, and mortality rates. It was estimated that direct medical expenses for those diagnosed with diabetes in Alabama were about $4.2 billion in 2021 (American Diabetes Association, 2021). Due to the overall burden of the disease, there has been an increased focus on developing innovative strategies such as community-based interventions and diabetes education. The project aims to improve participation, retention, engagement, and clinical outcomes (HbA1C) of adults aged 18 and over living with diabetes in Jefferson County, Alabama in diabetes self-management education and support programs where the population lives, works, and plays. Leveraging a dynamic, multi-directional recruitment model through a collaborative partnership with community health workers (CHWs) and local primary care providers and a diabetes-related mobile application, the investigators plan to test, via a randomized controlled trial (RCT), the combined effects of a community health worker-led, muli-directional recruitment process versus a traditional recruiting process involving flyers, word-of-mouth, and media ads. The investigators also propose to assess the effectiveness of adding a diabetes-related mobile application (HICO Health) that, through a user-friendly interface, allows patients to review on-demand, evidence-based videos, nutrition education, and behavior change surveys to supplement standard DSMES curriculum, as well as a tool to collect patient entered clinical data such as blood pressure and blood sugar readings. The HICO Health package also includes a provider dashboard that allows the diabetes care team to monitor, in real-time, patient clinical data as well as communicate to patients via the HIPAA-compliant messaging function. The specific aims of the study are as follows: Aim 1: To examine the effectiveness of utilizing a multi-directional recruitment model involving community health workers and primary care providers versus traditional recruitment methods (including using flyers, word of mouth, and media ads) to recruit people living with diabetes into a pharmacist-led DSMES program. Aim 2: To conduct a pilot/feasibility study comparing using the HICO Health app as a supplement to a standard DSMES curriculum to improve patient participation, retention, and patient clinical outcomes in a pharmacist-led DSMES program versus the standard DSMES alone in Jefferson County, AL. Throughout the project, the study team and the diabetes care team will frequently communicate with the study stakeholders to seek input on relevant aspects of the study such as the engagement of CHWs, the stakeholders' perspective on the recruitment process, the number of participants referred and enrolled, and the clinical outcomes of the participants, to name a few. The evidence from the study will play a crucial role in establishing scalable and sustainable DSMES recruitment and delivery models to not only increase accessibility, participation, and retention in DSMES programs but also improve clinical outcomes in people living with diabetes in Jefferson County.

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident of Jefferson County, Alabama
* Must have an ICD-10 diagnosis of diabetes
* Must have a primary care provider
* Must be able to read, write, and converse in English
* Must own and be able to utilize a smartphone with internet access
* Must be willing to visit MedsPLUS Consulting in downtown Birmingham on 3 separate occasions (transportation may be provided, if approved).
* Must be willing to attend and participate in five, two-hour education sessions over the course of 10 weeks

Exclusion Criteria:

* Currently enrolled in a diabetes-related study
* Currently enrolled in a lifestyle change program
* Does not have or cannot get access to a home blood glucose monitor
* Does not have or cannot get access to a smartphone with internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of Referrals from Study Stakeholders | 3 months
  Number of referrals from study stakeholders to DSMES programs in Jefferson County, AL.
Number of Participants Enrolled in DSMES Study | 3 months
  Number of Participants Enrolled in DSMES Study
Number of DSMES Sessions Attended by Participants | 2 months
  Number of DSMES sessions attended
Number of DSMES Participants with at Least 80% Session Retention | 2 months
  Number of participants completing 4 of 5 DSMES sessions
Change in HbA1C of Participants | Baseline, 3 months, and 6 months
  Change in HbA1C

SECONDARY OUTCOMES:
Change in Self-Care Knowledge | 6 months
  Measure change in diabetes self-care knowledge utilizing the Diabetes Self-Management Questionnaire a 16-question survey broken down into 4 sub-scales (glucose management, dietary control, physical activity, and healthcare use). The rating scale utilizes a 4-point Likert scale ranging from 0 to 3 (where 0 means it does not apply to the participant and 3 means it applies to the participant very much). For each sub-scale, the minimum score is zero and the maximum score is 10, and higher scores are indicative of better self-care. Additionally, there is one item that requires participants to rate their perceived self-care using the 4-point Likert scale indicated above.
App Engagement | 6 months
  Number of participants who used app at least two times a week during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dashauna M Ballard, PhD, MPH, Principal Investigator — Lister Hill Center for Health Policy University of Alabama at Birmingham; Pauline K Long, PharmD, Principal Investigator — MedsPLUS Consulting LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adam L, O'Connor C, Garcia AC. Evaluating the Impact of Diabetes Self-Management Education Methods on Knowledge, Attitudes and Behaviours of Adult Patients With Type 2 Diabetes Mellitus. Can J Diabetes. 2018 Oct;42(5):470-477.e2. doi: 10.1016/j.jcjd.2017.11.003. Epub 2017 Nov 23. PMID 29449096
- [Background] Adu MD, Malabu UH, Malau-Aduli AEO, Malau-Aduli BS. Users' preferences and design recommendations to promote engagements with mobile apps for diabetes self-management: Multi-national perspectives. PLoS One. 2018 Dec 10;13(12):e0208942. doi: 10.1371/journal.pone.0208942. eCollection 2018. PMID 30532235
- [Background] Alabama Department of Public Health. (2020). Diabetes. Available at https://www.alabamapublichealth.gov/healthrankings/assets/2020_sha_health_indicator_13.pdf. Accessed on [August 14, 2022].
- [Background] Alcantara-Aragon V. Improving patient self-care using diabetes technologies. Ther Adv Endocrinol Metab. 2019 Jan 28;10:2042018818824215. doi: 10.1177/2042018818824215. eCollection 2019. PMID 30728941
- [Background] American Association of Diabetes Educators (2014). Competencies for diabetes educators. Available at https://www.diabeteseducator.org/docs/default-source/legacy-docs/_resources/pdf/general/comp002.pdf?sfvrsn=9. Accessed on [August 10, 2022].
- [Background] American Diabetes Association. (2021). The burden of diabetes in Alabama. Available at https://diabetes.org/sites/default/files/2021-10/ADV_2021_State_Fact_sheets_Alabama.pdf. Accessed on [August 14, 2022].
- [Background] Adjei Boakye E, Varble A, Rojek R, Peavler O, Trainer AK, Osazuwa-Peters N, Hinyard L. Sociodemographic Factors Associated With Engagement in Diabetes Self-management Education Among People With Diabetes in the United States. Public Health Rep. 2018 Nov;133(6):685-691. doi: 10.1177/0033354918794935. Epub 2018 Sep 17. PMID 30223759
- [Background] Centers for Disease Control and Prevention. (2021). Diabetes self-management education. Available at https://www.cdc.gov/diabetes/dsmes-toolkit/standards/index.html. Accessed on [August 14, 2022].
- [Background] Chatterjee S, Davies MJ, Heller S, Speight J, Snoek FJ, Khunti K. Diabetes structured self-management education programmes: a narrative review and current innovations. Lancet Diabetes Endocrinol. 2018 Feb;6(2):130-142. doi: 10.1016/S2213-8587(17)30239-5. Epub 2017 Sep 29. PMID 28970034
- [Background] Kavookjian J, LaManna JB, Davidson P, Davis JW, Fahim SM, McDaniel CC, Ekong G, Todd A, Yehl K, Cox C. Impact of Diabetes Self-Management Education/Support on Self-Reported Quality of Life in Youth With Type 1 or Type 2 Diabetes. Sci Diabetes Self Manag Care. 2022 Oct;48(5):406-436. doi: 10.1177/26350106221115450. Epub 2022 Jul 28. PMID 35899815
- [Background] Chrvala CA, Sherr D, Lipman RD. Diabetes self-management education for adults with type 2 diabetes mellitus: A systematic review of the effect on glycemic control. Patient Educ Couns. 2016 Jun;99(6):926-43. doi: 10.1016/j.pec.2015.11.003. Epub 2015 Nov 22. PMID 26658704
- [Background] Hunt CW. Technology and diabetes self-management: An integrative review. World J Diabetes. 2015 Mar 15;6(2):225-33. doi: 10.4239/wjd.v6.i2.225. PMID 25789104
- [Background] Hildebrand JA, Billimek J, Olshansky EF, Sorkin DH, Lee JA, Evangelista LS. Facilitators and barriers to research participation: perspectives of Latinos with type 2 diabetes. Eur J Cardiovasc Nurs. 2018 Dec;17(8):737-741. doi: 10.1177/1474515118780895. Epub 2018 Jun 11. PMID 29886773
- [Background] Krall JS, Kanter JE, Ruppert KM, Arena VC, Solano FX, Siminerio LM. Effect of a Primary Care-Based Diabetes Education Model on Provider Referrals and Patient Participation. Sci Diabetes Self Manag Care. 2021 Feb;47(1):74-84. doi: 10.1177/0145721720981840. PMID 34078203
- [Background] Narindrarangkura P, Boren SA, Khan U, Day M, Simoes EJ, Kim MS. SEE-Diabetes, a patient-centered diabetes self-management education and support for older adults: Findings and information needs from patients' perspectives. Prim Care Diabetes. 2022 Jun;16(3):395-403. doi: 10.1016/j.pcd.2022.02.008. Epub 2022 Feb 25. PMID 35227635
- [Background] Olesen K, Folmann Hempler N, Drejer S, Valeur Baumgarten S, Stenov V. Impact of patient-centred diabetes self-management education targeting people with type 2 diabetes: an integrative review. Diabet Med. 2020 Jun;37(6):909-923. doi: 10.1111/dme.14284. Epub 2020 Mar 20. PMID 32124483
- [Background] Powers MA, Bardsley J, Cypress M, Duker P, Funnell MM, Hess Fischl A, Maryniuk MD, Siminerio L, Vivian E. Diabetes Self-management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. Diabetes Care. 2015 Jul;38(7):1372-82. doi: 10.2337/dc15-0730. Epub 2015 Jun 5. No abstract available. PMID 26048904
- [Background] Shirvani T, Javadivala Z, Azimi S, Shaghaghi A, Fathifar Z, Devender Bhalla HDR, Abdekhoda M, Nadrian H. Community-based educational interventions for prevention of type II diabetes: a global systematic review and meta-analysis. Syst Rev. 2021 Mar 20;10(1):81. doi: 10.1186/s13643-021-01619-3. PMID 33743839
- [Background] Siminerio, L. M., Ruppert, K., Emerson, S., Solano, F. X., & Piatt, G. A. (2008). Delivering diabetes self-management education (DSME) in primary care: the Pittsburgh regional initiative for diabetes education (PRIDE). Disease Management & Health Outcomes, 16, 267-272.
- [Background] UAB Medicine. (2019). Community Health Needs Assessment. Available at https://www.uabmedicine.org/documents/142028/185199/CHNA+UAB+2019_FINAL+Approved.pdf/0634e584-3ac6-fdb9-9262-5f33c4a0cbdd. Accessed on [August 14, 2022].
- [Background] US Census Bureau. (2022a). Quick facts: Birmingham city. Available at https://www.census.gov/quickfacts/birminghamcityalabama. Accessed on [June 22, 2023].
- [Background] US Census Bureau. (2022b). Quick facts: Jefferson County. Available at https://www.census.gov/quickfacts/jeffersoncountyalabama. Accessed on [June 22, 2023].
- [Background] Schmitt A, Gahr A, Hermanns N, Kulzer B, Huber J, Haak T. The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control. Health Qual Life Outcomes. 2013 Aug 13;11:138. doi: 10.1186/1477-7525-11-138. PMID 23937988